CLINICAL TRIAL: NCT04388527
Title: An Open-Label, Single Arm, Phase 1, Safety and Exploratory Efficacy Study of Convalescent Plasma for Severely Ill Mechanically Ventilated Participants With COVID-19 Caused by SARS-CoV-2
Brief Title: COVID-19 Convalescent Plasma for Mechanically Ventilated Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 842996 (PennCCP-01)
Record Dates: First submitted 2020-05-04; First posted 2020-05-14 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Penn COVID-19 convalescent plasma
  Interventions: Biological: COVID-19 Convalescent Plasma

INTERVENTIONS:
Biological: COVID-19 Convalescent Plasma — Participants will receive 2 units of convalescent plasma collected from ABO-compatible donors who have recovered from COVID-19.

SUMMARY:
The purpose of this study is to see if this plasma can be safely used in humans with COVID-19 and to see if it can improve patients' health when they are sick with COVID-19.

DETAILED DESCRIPTION:
This open-label, single arm, phase 1 trial will assess the safety and efficacy of convalescent plasma in severely ill, mechanically ventilated participants with pneumonia due to COVID-19. This study will enroll adults 18 years old and older, including pregnant women. A total of 50 eligible participants will receive 2 units of convalescent plasma collected from ABO-compatible donors who have recovered from COVID-19. Participants will receive convalescent plasma on Study Day 1 in addition to standard of care. Participants will be assessed daily while hospitalized and then on Study Days 15, 22, 29, and 60. All participants will undergo a series of safety, efficacy, and laboratory assessments. Blood samples will be collected on Days 1 (prior to plasma administration), 3, 5, 8, 11, 15, 29, and 60. Oropharyngeal or endotracheal samples will be collected on Days 1 (prior to plasma administration), 3, 5, 8, 11, and 15.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years of age
2. Laboratory-confirmed SARS-CoV-2 infection as determined by PCR or other authorized or approved assay in any specimen collected within 72 hours prior to enrollment. Note - An exception must be requested to the Sponsor if≥72 hours since positive test.
3. Hospitalized, on invasive mechanical ventilation or ECMO, consistent with a clinical status assessment 8-point ordinal scale severity score of 7.
4. Documentation of pneumonia with radiographic evidence of infiltrates by imaging (e.g., chest x-ray or CT scan).
5. Patient or proxy is willing and able to provide written informed consent and comply with all protocol requirements.

Exclusion Criteria:

1. Contraindication to transfusion (e.g., severe volume overload, history of severe allergic reaction to blood products), as judged by the investigator.
2. Clinical suspicion that the etiology of acute illness (acute decompensation) is primarily due to a condition other than COVID-19
3. Receipt of other investigational therapy as a part of another clinical trial. a. Note: investigational therapies used as part of clinical care, (eg, remdesivir, hydroxychloroquine) are permissible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine J. Bar, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 32
Completed | 15
Not Completed | 17
Not completed — Death | 14
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 10
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Participants With Serious Adverse Events.
Description: Cumulative incidence of participants with at least one serious adverse events (SAEs) at Study Day 29.
Time Frame: Up to Study Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 32
Participants | 22

2. Primary Outcome: Time to Clinical Improvement.
Description: Time to removal from mechanical ventilation.
Time Frame: Up to Study Day 29
Population: excludes those without improvement (were still on mechanical ventilation or died before removal of invasive mechanical ventilation/ECMO)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment
Number analyzed (Participants) | 15
Days | 11 [5 to 15.5]

3. Secondary Outcome: Clinical Status Assessment, Using 8-point Ordinal Scale, of Convalescent Plasma Administration
Description: Time to improvement by at least 2 category from Day 1 (time to reach WHO8 <=5). WHO8 score:
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities and/or requiring home oxygen;
  3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care;
  4. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise);
  5. Hospitalized, requiring supplemental oxygen;
  6. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  7. Hospitalized, on invasive mechanical ventilation or ECMO;
  8. Death
Time Frame: Up to Study Day 29
Population: excludes those without improvement (WHO8 score of 6,7,or 8)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 12
days | 12.5 [6 to 16.25]

4. Secondary Outcome: Clinical Status Assessment Using the National Early Warning Score (NEWS) of Convalescent Plasma Administration
Description: Time to discharge or to a NEWS of ≤ 2 and maintained for 24 hours, whichever occurs first.
  NEWS assessed daily while hospitalized until discharge or death and on Days 15 and 29.
  Higher NEWS is worse, range from 0 to 20.
Time Frame: Up to Study Day 29
Population: excludes 20 subjects who have outcome measure of Infinity as they were never discharged or never had NEWS <=2 while in hospital by Study Day 29
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 12
days | 10 [6 to 17.5]

5. Secondary Outcome: Incidence of New Oxygenation Use up to Day 29 of Convalescent Plasma Administration
Description: Incidence of new oxygenation use up to Day 29.
Time Frame: From enrollment to Day 29.
Population: this endpoint was not measured due to redundancy
Arm/Group | Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of New Oxygen Use up to Day 29 of Convalescent Plasma Administration
Description: Days of new oxygen use up to Day 29.
Time Frame: From enrollment to Day 29.
Population: this endpoint was not measured due to redundancy
Arm/Group | Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Oxygenation
Description: Days of supplemental oxygen while in hospital up to Study Day 29. In hospital supplemental oxygen days counted as days with a WHO8 ordinal score of 5, 6, or 7.
Time Frame: Daily while hospitalized up to Study Day 29.
Population: All 32 enrolled subjects were evaluated for days of oxygenation.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 32
days | 16 [7 to 23]

8. Secondary Outcome: Non-invasive Ventilation/High Flow Oxygen Days up to Day 29 of Convalescent Plasma Administration.
Description: Days of non-invasive ventilation/high flow oxygen while in hospital up to Day 29, defined as having WHO8 ordinal score of 6 = Hospitalized, on non-invasive ventilation or high flow oxygen devices
Time Frame: Daily while in hospital to Study Day 29.
Population: All 32 enrolled subjects were evaluated. Subjects who never had a WHO8 ordinal score of 6 = Hospitalized, on non-invasive ventilation or high flow oxygen devices have a measured outcome of 0 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 32
days | 0 [0 to 2]

9. Secondary Outcome: Number of Subjects With at Least One Day of Non-invasive Ventilation/High Flow Oxygen up to Day 29 of Convalescent Plasma Administration.
Description: Number of subjects with at least one day of non-invasive ventilation (WHO8 ordinal score of 6) while in hospital
Time Frame: Daily while in hospital to Study Day 29.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 32
Participants | 13

10. Secondary Outcome: Duration of Non-invasive Ventilation/High Flow Oxygen up to Day 29 of Convalescent Plasma Administration.
Description: Days of non-invasive ventilation/high flow oxygen up to Day 29.
Time Frame: Daily while in hospital to Study Day 29.
Population: this endpoint was not measured due to redundancy with other endpoints (#8)
Arm/Group | Treatment
Number analyzed (Participants) | 0

11. Secondary Outcome: Invasive Ventilation/ Extracorporeal Membrane Oxygenation(ECMO) Days
Description: Days on Invasive Ventilator/ECMO defined as WHO8 ordinal score of 7 = Hospitalized, on invasive mechanical ventilation or ECMO
Time Frame: Daily while in hospital to Study Day 29
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 32
days | 11.5 [5.75 to 19.25]

12. Secondary Outcome: Incidence of New Mechanical Ventilation or ECMO Use of Convalescent Plasma Administration.
Description: Incidence of new mechanical ventilation or ECMO use up to Day 29.
Time Frame: From enrollment to Day 29.
Population: Endpoint was not well defined as all subjects started on mechanical ventilation
Arm/Group | Treatment
Number analyzed (Participants) | 0

13. Secondary Outcome: Duration of New Mechanical Ventilation or ECMO Use of Convalescent Plasma Administration.
Description: Days of new mechanical ventilation or ECMO use up to Day 29.
Time Frame: From enrollment to Day 29.
Population: Endpoint was not well defined as all subjects started on mechanical ventilation
Arm/Group | Treatment
Number analyzed (Participants) | 0

14. Secondary Outcome: Duration of Hospitalization
Description: Duration (days) of first hospitalization. Time until death or discharge or Study Day 29
Time Frame: To Study Day 29
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 32
days | 20 [9.5 to 26.5]

15. Secondary Outcome: Mortality
Description: 28 day mortality
Time Frame: 28 days from Study Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 32
Participants | 14

16. Secondary Outcome: Serious Adverse Events (SAEs) Through Day 29 of Convalescent Plasma Administration.
Description: subjects with Serious Adverse Events (SAEs) through Day 29.
Time Frame: Through Study Day 29.
Population: .this endpoint is redundant with the primary endpoint
Arm/Group | Treatment
Number analyzed (Participants) | 0

17. Secondary Outcome: Number of Subjects With at Least One Grade 3 and Grade 4 Clinical and/or Laboratory Adverse Events Through Day 29 of Convalescent Plasma Administration.
Description: Number of subjects with at least one Grade 3 or Grade 4 clinical and/or laboratory adverse events through Day 29.
Time Frame: Through Study Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 32
Participants | 32

18. Secondary Outcome: Changes in WBC With Differential Through Day 29 of Convalescent Plasma Administration.
Description: Collected labs on Days 1 (baseline), 3, 5, 8, and 11 (while hospitalized), Days 15 and 29 (if attends in person visit or still hospitalized). Changes measured as difference between last measured lab value and baseline lab value. A negative value indicates last lab value > baseline lab value.
Time Frame: Through Day 29.
Population: Defined changes as difference between last measured lab value and baseline (day 1) lab value. Day of last measured lab may differ among subjects.
Measure: Median (Inter-Quartile Range); unit: THO/uL
Arm/Group | Treatment
Number analyzed (Participants) | 32
THO/uL | 1.25 [-4.40 to 7.00]

19. Secondary Outcome: Changes in Hemoglobin Measurement Through Day 29 of Convalescent Plasma Administration.
Description: as for outcome 18
Time Frame: Through Day 29.
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Treatment
Number analyzed (Participants) | 32
g/dL | -0.65 [-2.40 to 0.475]

20. Secondary Outcome: Changes in Platelets Measurement Through Day 29 of Convalescent Plasma Administration.
Description: as for outcome 18
Time Frame: Through Day 29.
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: 10^3 platelets per uL
Arm/Group | Treatment
Number analyzed (Participants) | 32
10^3 platelets per uL | 24 [-105.75 to 90.00]

21. Secondary Outcome: Changes in Creatinine Measurement Through Day 29 of Convalescent Plasma Administration.
Description: as for outcome 18
Time Frame: Through Day 29.
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 32
mg/dL | -0.39 [-1.505 to -0.010]

22. Secondary Outcome: Changes in Glucose Measurement Through Day 29 of Convalescent Plasma Administration.
Description: as for outcome 18
Time Frame: Through Day 29.
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 32
mg/dL | -36.00 [-81.50 to -2.25]

23. Secondary Outcome: Changes in Total Bilirubin Measurement Through Day 29 of Convalescent Plasma Administration.
Description: as for outcome 18
Time Frame: Through Day 29.
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 32
mg/dL | 0.00 [-0.100 to 0.225]

24. Secondary Outcome: Changes in ALT Measurement Through Day 29 of Convalescent Plasma Administration.
Description: as for outcome 18
Time Frame: Through Day 29.
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Treatment
Number analyzed (Participants) | 32
U/L | -3.00 [-20.25 to 17.50]

25. Secondary Outcome: Changes in AST Measurement Through Day 29 of Convalescent Plasma Administration.
Description: as for outcome 18
Time Frame: Through Day 29
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Treatment
Number analyzed (Participants) | 32
U/L | -7.50 [-33.00 to 1.75]

26. Secondary Outcome: Changes in PT Measurement Through Day 29 of Convalescent Plasma Administration.
Description: as for outcome 18
Time Frame: Through Day 29
Population: Defined changes as difference between last measured lab value and baseline (day 1) lab value. Day of last measured lab may differ among subjects.
  analyzed sample size is 30 because 2 subjects did not have PT lab collected.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Treatment
Number analyzed (Participants) | 30
seconds | -0.050 [-2.950 to 1.075]

ADVERSE EVENTS:
Time Frame: Up to 65 days after receiving investigational product
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 14/32
Serious Adverse Events (participants affected / at risk) | 23/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=32)
Acute CNS Ischemia (Nervous system disorders) | 2 (2) — Cerebral vascular accident (e.g., stroke with neurological deficit)
Acidosis (Metabolism and nutrition disorders) | 1 (1) — Laboratory Value: Chemistries
Arrhythmia (by ECG or physical examination) (Cardiac disorders) | 2 (2) — Life-threatening arrhythmia OR Urgent intervention indicated
Creatinine Clearance Low (Renal and urinary disorders) | 1 (1)
Dyspnea or Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 13 (16)
Hemorrhage (with significant acute blood loss) (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 6 (6)
Embolism (Vascular disorders) | 1 (1) — Life-threatening embolic event (e.g., pulmonary embolism, thrombus)
Altered mental status (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=32)
Acidosis (Metabolism and nutrition disorders) | 9 (13)
Albumin, Low (Metabolism and nutrition disorders) | 5 (6)
Alkalosis (Metabolism and nutrition disorders) | 4 (5)
ALT, High (Investigations) | 3 (4)
Altered Mental Status (Nervous system disorders) | 5 (5)
Arrhythmia (Cardiac disorders) | 13 (19)
AST, High (Investigations) | 3 (3)
Blood Pressure Abnormalities Hypertension (with the lowest reading taken after repeat testing durin (Vascular disorders) | 8 (14)
Calcium, Low (Metabolism and nutrition disorders) | 4 (6)
Creatinine, High (Investigations) | 7 (9)
Fever (non-axillary temperatures only) (General disorders) | 7 (8)
Glucose (mg/dL; mmol/L) Fasting, High (Metabolism and nutrition disorders) | 8 (8)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemoglobin, Low (g/dL; mmol/L) >= 13 years of age (female only) (Blood and lymphatic system disorders) | 10 (14)
Hypotension (Vascular disorders) | 8 (13)
Lactate, High (Investigations) | 2 (2)
Platelets, Decreased (Blood and lymphatic system disorders) | 6 (8)
Sodium, High (Metabolism and nutrition disorders) | 7 (10)
Thrombosis or Embolism (Vascular disorders) | 4 (5)
Hemorrhage (with significant acute blood loss) (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin, Low (g/dL; mmol/L) >= 13 years of age (male only) (Blood and lymphatic system disorders) | 20 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT04388527/Prot_SAP_000.pdf